CLINICAL TRIAL: NCT05927766
Title: Correlation Between Endoscopic Findings And Helicobacter Pylori Infection In Chronic Kidney Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Faisal Abdellah, Principal investigator, Sohag University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: CKD and H.Pylori infection
Record Dates: First submitted 2023-05-12; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with chronic kidney disease (Active Comparator)
  Interventions: Device: esophagogastroduodenoscopy
- patients without chronic kidneys disease (Active Comparator)
  Interventions: Device: esophagogastroduodenoscopy

INTERVENTIONS:
Device: esophagogastroduodenoscopy — patients with upper gastrointestinal symptoms will gone to upper endoscopy and biopsy when indicated

SUMMARY:
The aim of this study is to

1. Evaluate frequency of H. pylori infection in patients with CKD.
2. Description the gastroduodenal lesions found in patients with chronic kidney disease and correlate it to H.pylori infection.

DETAILED DESCRIPTION:
cross sectional study to study the relationship between Helicobacter Pylori Infection and Gastroduodenal Lesions in Patients with Chronic Kidney Disease, There have been some debates about the association of Helicobacter pylori infection and chronic kidney disease (CKD). Pathogenesis of H. pylori infection in patients with CKD is not clearly revealed and there are not enough studies about these two factors.

There are several hypothesis which support that kidney disease may reduce H. pylori infection. High level of serum urea nitrogen can contribute to a decreased gastric acid secretion and higher gastric alkalosis which could be the cause of lower prevalence of H. pylori among CKD. Inflammatory cytokines are also increased in CKD patients and it can cause gastric mucosal damage, chronic gastritis, and spontaneously eradicate H. pylori. In addition, antibiotics, proton pump inhibitors, or H2 receptor antagonists which are used in patients with CKD for long time might be associated with decreased H. pylori infection.

There are other hypothesis that are contrary to above theories. Some studies showed that high u rea concentration makes the gastric mucosa more susceptible to H. pylori and infection rate is higher in uremic patients. And, in some articles which have studied about peptic ulcer in CKD, the prevalence of H. pylori infection looked lower compare to ulcer in non-CKD patients but real incidence may not be lower. Because the incidence of peptic ulcer is higher in CKD patients with various causes except H. pylori infection.

Gastrointestinal (GI) disorders are the most prevalent chronic problem in CKD patients, ranking second in frequency only to renal failure itself. GI disorders affect 70 to 80% of patients on Hemodialysis (HD); yet, little is known about the impact of Hp infection on this multifactorial disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD classified as stages 3 to 5 according Kidney Disease Improving Global Outcomes classification, on hemodialysis or not.
* control group without chronic kidney disease.

Exclusion Criteria:

* frail patients with multiple comorbidities or malignant disease.
* pregnant ladies.
* patients recently on proton pump inhibitors two weeks or less prior to the interview.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Description the gastroduodenal lesions found in upper endoscopy in patients with chronic kidney disease or not and correlate them to helicobacter pylori infection | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Usama a arafa, Study Director — Sohag University
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided